CLINICAL TRIAL: NCT04739202
Title: An Umbrella Phase 2 Trial to Assess Personalized Targeted IMMUNOtherapy-based Regimens in Recurrent Advanced/Metastatic GASTric Adenocarcinoma Patients
Brief Title: Personalized Targeted IMMUNOtherapy-based Regimens in Recurrent GASTric Adenocarcinoma (IMMUNOGAST)
Acronym: IMMUNOGAST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0153; 2020-000297-17 (EudraCT Number)
Record Dates: First submitted 2021-01-13; First posted 2021-02-04 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Gastric Adenocarcinoma; Metastatic Gastric Cancer; Metastatic Adenocarcinoma; Advanced Gastric Carcinoma
Keywords: Atezolizumab; Bevacizumab; Ipatasertib; Gastric adenocarcinoma; Umbrella phase 2 trial; Genomic landscape; Personalized Immunotherapy
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — atezolizumab; ipatasertib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with tumors positive for EBV or microsatellite instable tumors (group 1) (Experimental): Atezolizumab IV (1200 mg every 3 weeks) + Ipatasertib tablet (400 mg a day continuously).
  Interventions: Drug: Atezolizumab + Ipatasertib
- Patients with genomically stable tumors (group 2) (Experimental): Atezolizumab IV (1200 mg every 3 weeks) + Bevacizumab IV (15 mg/kg every 3 weeks).
  Interventions: Drug: Atezolizumab + Bevacizumab
- Patients with tumors with chromosomal instability (group 3) (Experimental): Atezolizumab IV (1200 mg every 3 weeks) + Bevacizumab IV (15 mg/kg every 3 weeks).
  Interventions: Drug: Atezolizumab + Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab + Ipatasertib — Atezolizumab IV (1200 mg on day 1 of each 21-day cycle) and Ipatasertib PO (400 mg per day continuously, starting on cycle 1 day 1). Treatment given until disease progression or unacceptable toxicity.
  Arms: Patients with tumors positive for EBV or microsatellite instable tumors (group 1)
Drug: Atezolizumab + Bevacizumab — Atezolizumab IV (1200 mg on day 1 of each 21-day cycle) and Bevacizumab IV (15 mg/kg on day 1 of each 21-day cycle). Treatment given until disease progression or unacceptable toxicity.
  Arms: Patients with genomically stable tumors (group 2); Patients with tumors with chromosomal instability (group 3)

SUMMARY:
For patients with advanced/metastatic gastric adenocarcinomas in progression after a first line chemotherapy comprising platinum and fluoropyrimidine, the reported second line treatments are : 1) paclitaxel combined with ramucirumab (overall response rate (ORR) = 25%; median progression free survival (PFS) = 2.9 months; median overall survival (OS)= 5.9 months), or paclitaxel alone (ORR = 14%, median PFS = 2.9 months; median OS= 5.9 months); 2) docetaxel (ORR = 7%, median OS = 5.2 months) or 3) irinotecan (ORR = 0%, median OS= 4.0 months).

These numbers demonstrate the poor prognosis of this disease, and the unmet medical need for innovative therapeutic strategies.

Cancer Genome Atlas (TCGA) mapped a genomic landscape of gastric adenocarcinomas, and identified 4 sub-types:

* Tumor positive for Epstein-Barr virus (EBV) (8%), which display recurrent PIK3CA mutations, extreme DNA hypermethylation, and amplification of JAK2, ErbB2, PD-L1 and PD-L2;
* Microsatellite instable tumors (MSI-high) (22%), which show elevated mutation rates, including mutations of genes encoding targetable oncogenic signaling proteins (PIK3CA, ErbB2, ErbB3, and EGFR);
* Genomically stable tumors (20%), which are enriched for the diffuse histological variant and mutations of RHOA or fusions involving RHO-family GTPase-activating proteins;
* Tumors with chromosomal instability (50%), which show marked aneuploidy and focal amplification of receptor tyrosine kinases and VEGFA.

Most of diffuse-type gastric adenocarcinomas were classified in genomically stable tumors. This subgroup of cancers, accounting for about 20 to 30% of gastric adenocarcinomas, is associated with particularly poor prognosis and resistance to chemotherapy. A proteomic landscape of diffuse-type gastric adenocarcinomas was recently reported.

Pembrolizumab, an anti-PDL1 drug granted with an accelerated approval by FDA in September 2017, exhibited promising activity in gastric adenocarcinoma patients previously treated with 1 or 2 lines of chemotherapy (ORR=11.6%, median PFS = 2.0 months, median OS= 5.6 months), especially in those with PDL1 positive tumors (ORR=22.7%). The tumor response was particularly high in patients with MSI-high tumor (ORR=57.1%). However the preliminary outcomes of the phase III KEYNOTE-061 trial (NCT02370498) recently released in the press suggest that pembrolizumab was not superior to paclitaxel in 592 patients with advanced gastric or gastroesophageal junction adenocarcinoma whose disease progressed after first-line treatment with platinum and fluoropyrimidine doublet therapy (the hazard ratio (HR) for OS was 0.82 (95% confidence interval = 0.66-1.03; one sided P = .042) (http://www.ascopost.com/News/58377).

These outcomes suggest that, although being very promising, immunotherapy should be combined to other agents for being fully effective in gastric adenocarcinomas patients.

We propose a strategy based on molecular features to select the drugs that will be associated with atezolizumab, an anti-PDL1 drug, in patients with pre-treated advanced gastric adenocarcinomas:

* Patients with tumors positive for EBV or microsatellite instable tumors (30%) will be treated with atezolizumab and ipatasertib.
* Patients with genomically stable tumors (20%) will be treated with atezolizumab combined with bevacizumab.
* Patients with tumors with chromosomal instability (50%) will be treated with atezolizumab combined with bevacizumab.

Expected outcomes:

IMMUNOGAST trial will provide data about the clinical feasibility of biomolecular characterization of gastric adenocarcinomas for routine treatment adjustment. Moreover it should generate information about the relevance of adjusting combined immunotherapies based on molecular subtypes, in terms of clinical efficacy. Finally, translational research project outcomes should provide important data about relationships between efficacy and tumor immune gene spatial expression, along with tumor and circulating mutational burden. These outcomes may help identify the best candidates for tested combinations in the future.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically documented recurrent advanced/metastatic gastric or gastroesophageal junction adenocarcinomas* previously treated with a platinum and fluoropyrimidine-based regimen.

  * The gastric or gastroesophageal junction adenocarcinomas that overexpress HER2 should have previously been treated with trastuzumab, except in the case of contraindication.
* Patients older than 18 years
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Patients must have documented disease progression
* Patients who have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Accessible tumor lesion (primitive lesion or metastasis) for trial dedicated tumor biopsy.
* Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (echo) or multigated acquisition (MUGA) scan within 28 days before day 1 of treatment.
* Child-Pugh class A
* Patients must have normal organ and marrow function:

  * Absolute neutrophil count ≥ 1,500/μL, platelets ≥ 100,000/μL, hemoglobin ≥ 9 g/dL
  * Total bilirubin ≤ 1.5 ULN except subject with documented Gilbert's syndrome, AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN, Serum alkaline phosphatase ≤ 2.5 x ULN. Patients with bone metastases: alkaline phosphatase ≤ 5 x ULN.
  * Albumin > 2.5 mg/dL.
  * Glomerular filtration rate ≥ 60 mL/min as determined by the CKD-EPI equation (or reference methodology such as Iohexol or isotopic technic).
  * Urine dipstick for proteinuria < 2+. If urine dipstick is ≥ 2+, 24-hour urine must demonstrate < 1 g of protein in 24 hours.
  * Normal blood pressure or adequately treated and controlled hypertension (systolic BP ≤ 140 mmHg and/or diastolic BP ≤ 90 mmHg).
* Female patients of childbearing potential must have a negative serum pregnancy test within 8 days of initiating protocol therapy.
* Female patients of childbearing potential must agree to use contraceptive methods with a low failure rate (< 1% per year) during the treatment period and for 6 months after the last dose of study drugs.
* Male patients of childbearing potential must agree to use contraceptive methods with a low failure rate during the treatment period and for 6 months after the last dose of study drugs.
* Patient is capable of understanding and complying with the protocol and has signed the informed consent document.
* Patients affiliated to a social insurance regime.

Exclusion Criteria:

* Residual toxicity from previous treatment grade ≥1, except for alopecia or peripheral neuropathy grade ≤ 2
* Radiotherapy within 28 days before inclusion, except for palliative radiotherapy if patients recovered from all side effects
* Congenital risk of bleeding, or acquired coagulopathy, or curative anti-coagulant therapies (except for low molecular weight heparin).
* Active digestive bleeding within 3 months before inclusion
* Patients pretreated with one of the experimental drugs, other immune checkpoint inhibitor anti-cancer drugs (anti-PD1, anti-PDL1, anti-CTLA4, …), or with ramucirumab.
* Uncontrolled high cholesterol or triglyceride grade ≥ 2
* Uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, congestive heart failure-New York Heart Association Class III or IV, active ischemic heart disease, myocardial infarction within the previous six months, uncontrolled diabetes mellitus, gastric or duodenal ulceration diagnosed within the previous 6 months, chronic liver or renal disease, or severe malnutrition.
* Current peripheral neuropathy of Grade ≥ 3 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.5.0
* Active, second potentially life-threatening cancer
* Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS). Patient with a history of localized malignancy diagnosed over 5 years ago may be eligible provided he completed her adjuvant systemic therapy and remains free of recurrent or metastatic disease.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
* Major surgery within 28 days before cycle 1, day 1
* Active infection requiring iv antibiotics at day 1 of cycle 1
* Medical condition that requires chronic systemic steroid therapy or on any other form of immunosuppressive medication. For example, patients with autoimmune disease that requires systemic steroids or immunosuppression agents should be excluded. Replacement therapy (eg., thyroxine, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs, resulting in dyspnea at rest
* Patient is positive for the human immunodeficiency virus (HIV), HepBsAg, or HCV RNA.
* Live vaccine within 28 days of planned start of study therapy
* History of abdominal fistula, gastrointestinal perforation and/or intra-abdominal abscess within the previous 6 months
* History of Type I or Type II diabetes mellitus requiring insulin
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins or Chinese Hamster Ovary (CHO) cell proteins or loperamide drug or excipient
* Known hypersensitivity to any of the components of atezolizumab, bevacizumab or ipatasertib
* Participation in other interventional clinical research that may interfere with the experimental drugs efficacy
* History of severe or life-threatening skin adverse reaction on prior treatment with other immune-stimulatory anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-10-26 (Estimated); Study Completion 2023-10-26 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Through the expected duration of the treatment, an average of 27 weeks and a maximum of 2 years (estimated)
  Objective response rate, using iRECIST, defined as the percentage of patients experiencing a complete response or a partial response, as their best tumor responses during the whole treatment period

SECONDARY OUTCOMES:
Overall survival | From the date of inclusion (Day -28 to Day 0) to the date of death or to the end of the study or in a complementary study (to collect vital status and date of death, every 3 months for 5 years for patients alive at the end of the study
  The overall survival (OS) will be measured from the date of inclusion to the date of death or to the end of the study or in a complementary study (to collect vital status and date of death, every 3 months for 5 years for patients alive at the end of the study).
Progression-free survival | From the date of inclusion (Day -28 to Day 0) to the date of disease progression, or death or to the end of the study up to 52.5 months
  The progression-free survival (PFS) will be evaluated according to iRECIST criteria.
Safety, treatment-related adverse events | 100 days after the last experimental treatment
  Treatment-related adverse events are defined as the nature, number and grade of adverse events observed throughout the study and assessed using NCI-CTCAE v.5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit YOU, MD, Principal Investigator — Service d'Oncologie Médicale - Centre Hospitalier Lyon Sud
Locations (8):
- France (8):
  - Dijon - Centre Georges-Francois Leclerc, Dijon
  - Hcl - Hopital Edouard Herriot, Lyon
  - Aphm - Hopital La Timone, Marseille
  - Aphp - Hopital Saint-Louis, Paris
  - Aphp - Hopital Pitie Salpetriere, Paris
  - Bordeaux - Hopital Haut-Leveque, Pessac
  - Hcl - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Toulouse - Iuct Rangueil-Larrey, Toulouse